CLINICAL TRIAL: NCT06213662
Title: Effect of Botulinum Toxin Injection Guided by Ultrasound Combined With Balloon Localization on Cricopharyngeal Achalasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yuli Zhu, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-0296-001
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cricopharyngeal Achalasia; Dysphagia
Keywords: Botulinum Toxins
MeSH Terms: conditions — Deglutition Disorders | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Botulinum toxin type A for injection (Hengli National Drug approval number S10970037) 100U, diluted with
  1 ml.9% sodium chloride solution for reserve use.Each patient was injected with 90U
  Interventions: Drug: Botulinum toxin type A for injection

INTERVENTIONS:
Drug: Botulinum toxin type A for injection — Botulinum toxin was injected into the upper esophageal sphincter of each patient
  Other Names: Botulinum toxin type A for injection (Hengli National Drug approval number S10970037)

SUMMARY:
cricopharyngeal achalasia refers to incomplete or non-open functional opening of the cricopharyngeal muscle, and after repeated swallowing of food, it still cannot pass through the cricopharyngeal muscle, remaining in the epiglottic valley and the piriform fossa, and even regurgitated into the nasal cavity . Neurogenic diseases, myogenic diseases and head and neck tumors are the common causes. Patients with chronic underfeeding lead to malnutrition, reduced quality of life, affecting the outcome of the disease. At present, the treatment measures for cricopharyngeal achalasia at home and abroad include balloon dilation technique, surgical incision, botulinum toxin injection. The dilation of the balloon is easy to cause mucosal edema and damage. Local infection, massive hemorrhage, local nerve injury and other complications often occur in cricopharyngotomy. Botulinum toxin injection relieves muscle spasms and is now widely used to treat dystonia. Common injection localization methods include CT, ultrasound, electromyography and endoscopy. Ultrasound-guided injection is a new technique of visualization, simple and non-radiation injection guidance, which can observe the injection process and drug injection position in real time. Fixation with a balloon can further improve the accuracy of the injection. In this study, botulinum toxin was injected into the cricopharyngeal muscle by ultrasound combined with balloon.

DETAILED DESCRIPTION:
Under the ultrasound combined with balloon fixation, two injection sites were selected from the left upper esophageal sphincter, and 30U was injected respectively, and one injection site was selected from the right side, and 30U was injected. In addition, the patient also received routine swallowing training once a day for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The videofluoroscopic swallowing study (VFSS) confirmed that the cricopharyngeal muscle was not open/closed
* Patients with no significant improvement in swallowing function after more than 2 weeks of standardized rehabilitation therapy (FOIS unchanged or decreased)
* In the presence of swallowing initiation, VFSS is seen in swallowing with an upward motion of the hyoid greater than half the height of the C3 cone
* Vital signs stable, conscious, treatment cooperative
* The patient himself or his family members sign the written informed consent voluntarily

Exclusion Criteria:

* Patients with severe cognitive impairment, mental illness, and severe cardiopulmonary disease
* The structure of the throat is abnormal
* Malignant tumor patient
* Infection or wound at the injection site
* People allergic to botulinum toxin
* Bleeding tendency and coagulation disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale | pre-treatment、2 weeks after treatment、4 weeks after treatment、24 weeks after treatment
  According to whether the patient can eat by mouth and the degree of dependence on nasal feeding tube, it is divided into 7 grades, corresponding to 1-7 points respectively. The higher the score, the better the swallowing function.
Rosenbek penetration-aspiration scale | pre-treatment、2 weeks after treatment、4 weeks after treatment、24 weeks after treatment
  Based on the results of Videofluroscopic swallowing study (VFSS), the cases of leakage and aspiration were divided into 8 grades, corresponding to 1-8 points respectively. The higher the score, the better the swallowing function.

SECONDARY OUTCOMES:
Murray secretion scale | pre-treatment、2 weeks after treatment
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), the accumulation position of oropharyngeal secretions was described and divided into 4 grades. The higher the score, the worse the swallowing function.
yale pharyngeal residue severity rating scale | pre-treatment、2 weeks after treatment
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), the main indicators include the location of the residue (epiglottic valley and pyriform sinus) and the amount of residue, which is divided into 5 grades. The higher the score, the worse the swallowing function.
fiberoptic endoscopic dysphagia severity scale | pre-treatment、2 weeks after treatment
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), Eat different foods and observe whether penetration aspiration and protective reflex occur. The highest score is 6, which means that saliva accumulates with penetration or aspiration, and the lowest score is 1. When eating soft solid food, there is no leakage or aspiration, and there is little or moderate residue in epiglottic valley or pyriform sinus. The higher the score, the worse the swallowing function.

CONTACTS AND LOCATIONS:
Overall Officials: Yuli Zhu, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No
Due to the privacy policy of the First Affiliated Hospital of Zhengzhou University,the data cannot be disclosed, but it can be obtained from the PI with an appropriate reason